CLINICAL TRIAL: NCT00044733
Title: A Dose-Finding Study of the Safety of Gemtuzumab Ozogamicin as Single Agent Treatment of Patients With Relapsed Acute Myelogenous Leukemia After Autologous or Allogenic Hematopoietic Stem Cell Transplant (HSCT)
Brief Title: Study Evaluating Gemtuzumab Ozogamicin in Acute Myelogenous Leukemia After Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Masking: None
Other Study IDs: 0903X-100374; NCT00053274 (obsolete NCT alias)
Record Dates: First submitted 2002-09-04; First posted 2002-09-06 (Estimated); Last update posted 2006-05-18 (Estimated); Status verified 2006-05

CONDITIONS: Acute Myelogenous Leukemia
Keywords: Leukemia; Stem Cell Transplant
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — Gemtuzumab; Injections

INTERVENTIONS:
Drug: Mylotarg (gemtuzumab ozogamicin) Injection

SUMMARY:
The primary objective of this study is to evaluate the safety of gemtuzumab ozogamicin in relapsed CD33-positive AML patients who received HSCT. If the MTD dose is not reached, 9 mg/m2 will be the maximum tested dose. A secondary objective is to assess efficacy in terms of the number of patients attaining a complete (CR) or morphological (CRp) remission.

ELIGIBILITY:
Inclusion Criteria

* Patients with CD33+ AML who have experienced relapse after autologous or allogeneic HSCT. Flow cytometry, performed at the study site, must demonstrate that the patient has AML that is CD33 positive, based on local laboratory criteria (Patients with history of MDS pretransplant will be eligible if their proportion of myeloblasts by marrow aspirate exceeds 5% at time of evaluation for Gemtuzumab Ozogamicin treatment)
* The patient must be greater than or equal to 60 days post-HCST
* Patients of all ages may be entered in this study

Exclusion Criteria

* Peripheral white blood count (WBC) greater than or equal to 30,000/uL at the time of initial Gemtuzumab Ozogamicin administration. (In order to reduce the peripheral blood count, patients may be treated with Hydroxyurea. Hydroxyurea must be discontinued 24 hours prior to Gemtuzumab Ozogamicin administration.)
* Known active central nervous system (CNS) or testicular leukemia at time of study entry.
* Prior therapy with anti-CD33 antibodies.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38
Dates: Start 2000-03; Study Completion 2004-09

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (13):
- United States (13):
  - Little Rock, Arkansas
  - Hartford, Connecticut
  - Jacksonville, Florida
  - Honolulu, Hawaii
  - Olathe, Kansas
  - Camden, New Jersey
  - Trenton, New Jersey
  - Buffalo, New York
  - Rochester, New York
  - Canton, Ohio
  - Houston, Texas
  - Charleston, West Virginia
  - Madison, Wisconsin